CLINICAL TRIAL: NCT04410978
Title: A Phase 3, Randomized, Double-blind Efficacy and Safety Study Comparing SAR442168 to Teriflunomide (Aubagio®) in Participants With Relapsing Forms of Multiple Sclerosis
Brief Title: Relapsing Forms of Multiple Sclerosis (RMS) Study of Bruton's Tyrosine Kinase (BTK) Inhibitor Tolebrutinib (SAR442168) (GEMINI 1)
Acronym: GEMINI 1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: EFC16033; U1111-1238-1418 (Registry Identifier: ICTRP); 2020-000637-41 (EudraCT Number); NCT04964791 (obsolete NCT alias)
Record Dates: First submitted 2020-05-28; First posted 2020-06-01 (Actual); Results first posted 2025-06-18 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-06

CONDITIONS: Relapsing Multiple Sclerosis
MeSH Terms: interventions — teriflunomide

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- SAR442168 (Experimental): 60 mg oral SAR442168 + placebo to match the teriflunomide tablet once daily
  Interventions: Drug: Tolebrutinib; Drug: Placebo to match Teriflunomide
- Teriflunomide (Active Comparator): 14 mg oral teriflunomide + placebo to match the SAR442168 tablet once daily
  Interventions: Drug: Teriflunomide; Drug: Placebo to match Tolebrutinib

INTERVENTIONS:
Drug: Tolebrutinib — Pharmaceutical form: Tablet
  Route of administration: Oral
  Other Names: SAR442168
  Arms: SAR442168
Drug: Teriflunomide — Pharmaceutical form: Tablet
  Route of administration: Oral
  Arms: Teriflunomide
Drug: Placebo to match Tolebrutinib — Pharmaceutical form: Tablet
  Route of administration: Oral
  Arms: Teriflunomide
Drug: Placebo to match Teriflunomide — Pharmaceutical form: Tablet
  Route of administration: Oral
  Arms: SAR442168

SUMMARY:
Primary Objective:

To assess efficacy of daily SAR442168 compared to a daily dose of 14 mg teriflunomide (Aubagio) measured by annualized adjudicated relapse rate (ARR) in participants with relapsing forms of MS

Secondary Objective:

To assess efficacy of SAR442168 compared to teriflunomide (Aubagio) on disability progression, MRI lesions, cognitive performance and quality of life To evaluate the safety and tolerability of daily SAR442168 To evaluate population pharmacokinetics (PK) of SAR442168 and relevant metabolites and its relationship to efficacy and safety To evaluate pharmacodynamics (PD) of SAR442168

DETAILED DESCRIPTION:
This was an event-driven (6-month confirmed disability worsening [CDW]) trial with a variable treatment duration (end-of-study [EOS] duration: up to approximately 48 months).

ELIGIBILITY:
Inclusion criteria :

* The participant must be 18 to 55 years of age, inclusive, at the time of signing the informed consent
* The participant must have been diagnosed with RMS according to the 2017 revision of the McDonald diagnostic criteria
* The participant has an expanded disability status scale (EDSS) score ≤5.5 at the first Screening Visit
* The participant must have at least 1 of the following prior to screening:

  * ≥1 documented relapse within the previous year OR
  * ≥2 documented relapses within the previous 2 years, OR
  * ≥1 documented Gd enhancing lesion on an MRI scan within the previous year
* Contraceptive use by men or women should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies
* Male participants are eligible to participate if they agree to the following during the intervention period and until accelerated elimination procedure:

  * Refrain from donating sperm

Plus either:

* Be abstinent from heterosexual intercourse as their preferred and usual lifestyle (abstinent on a long term and persistent basis) and agree to remain abstinent OR
* Must agree to use contraception/barrier as detailed below:

Agree to use a male condom and should also be advised of the benefit for a female partner to use a highly effective method of contraception as a condom may break or leak when having sexual intercourse with a woman of childbearing potential (WOCBP) who is not currently pregnant

* A female participant is eligible to participate if she is not pregnant or breastfeeding, and at least one of the following conditions apply:

  * Is not a WOCBP OR
  * Is a WOCBP and agrees to use a contraceptive method that is highly effective (with a failure rate of <1% per year), preferably with low user dependency, during the intervention period and until accelerated elimination procedure is completed (or for at least 10 days after the last dose of SAR442168, if the case was unblinded)
* A WOCBP must have a negative highly sensitive pregnancy test at screening and within 24hours before the first dose of study intervention.
* If a urine test cannot be confirmed as negative (eg, an ambiguous result), a serum pregnancy test is required. In such cases, the participant must be excluded from participation if the serum pregnancy result is positive.
* The Investigator is responsible for review of medical history, menstrual history, and recent sexual activity to decrease the risk for inclusion of a woman with an early undetected pregnancy.
* The participant must have given written informed consent prior to undertaking any study related procedure. This includes consent to comply with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol. In countries where the legal age of maturity is greater than 18 years, a specific ICF for such legally minor participants must also be signed by the participant's legally authorized representative

Exclusion criteria:

* The participant has been diagnosed with primary progressive multiple sclerosis (PPMS) according to the 2017 revision of the McDonald diagnostic criteria or with nonrelapsing secondary progressive multiple sclerosis (SPMS)
* The participant has a history of infection or may be at risk for infection including but not limited to: HIV, transplantation, live attenuated vaccines, progressive multifocal leukoencephalopathy, tuberculosis, any persistent chronic or active recurring infection
* Clinically significant laboratory abnormalities (including evidence of liver injury) or electrocardiogram abnormalities at Screening.
* The participant has conditions or situations that would adversely affect participation in this study, including but not limited to:

  * A short life expectancy due to pre-existing health condition(s) as determined by their treating neurologist
  * Medical condition(s) or concomitant disease(s) making them nonevaluable for the primary efficacy endpoint or that would adversely affect participation in this study, as judged by the Investigator
  * A requirement for concomitant treatment that could bias the primary evaluation
* The participant has a history of or currently has concomitant medical or clinical conditions that would adversely affect participation in this study
* At screening, the participant is positive for hepatitis B surface antigen and/or hepatitis B core antibody and/or is positive for hepatitis C antibody
* The participant has any of the following:

  * A bleeding disorder or known platelet dysfunction at any time prior to the screening visit
  * A platelet count <150 000/μL at the screening visit
* The participant has a lymphocyte count below the lower limit of normal (LLN) at the screening visit
* The presence of psychiatric disturbance or substance abuse
* Prior/concomitant therapy
* The participant is receiving potent and moderate inducers of cytochrome P450 (CYP) 3A or potent inhibitors of CYP2C8 hepatic enzymes
* The participant is receiving anticoagulant/antiplatelet therapies

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 974 (Actual)
Dates: Start 2020-06-30 (Actual); Primary Completion 2024-07-15 (Actual); Study Completion 2024-07-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (179):
- United States (23):
  - University of Alabama MS Center-Site Number:8400013, Birmingham, Alabama
  - University of San Francisco, Sandler Neurosciences Center-Site Number:8400137, San Francisco, California
  - University of Colorado-Site Number:8400012, Aurora, Colorado
  - Georgetown University Medical Center-Site Number:8400119, Washington D.C., District of Columbia
  - Beth Israel Deaconess Medical Center-Site Number:8400064, Fort Myers, Florida
  - Axiom Clinical Research of Florida-Site Number:8400001, Tampa, Florida
  - University of South Florida-Site Number:8400006, Tampa, Florida
  - Meridian Clinical Research-Site Number:8400003, Savannah, Georgia
  - Consultants In Neurology-Site Number:8400011, Northbrook, Illinois
  - Tufts Medical Center-Site Number:8400072, Boston, Massachusetts
  - Michigan Institute For Neurological Disorders-Site Number:8400058, Farmington Hills, Michigan
  - The Memorial Hospital-Site Number:8400033, Owosso, Michigan
  - Sharlin Health & Neurology-Site Number:8400093, Ozark, Missouri
  - Missouri Baptist Medical Center-Site Number:8400019, St Louis, Missouri
  - Meridian Clinical Research, LLC-Site Number:8400005, Raleigh, North Carolina
  - Wake Forest University Baptist Medical Center-Site Number:8400116, Winston-Salem, North Carolina
  - The Ohio State University Wexner Medical Center-Site Number:8400150, Columbus, Ohio
  - Optimed Research, LTD-Site Number:8400147, Columbus, Ohio
  - Columbus Neuroscience-Site Number:8400010, Westerville, Ohio
  - Oklahoma Medical Research Foundation-Site Number:8400018, Oklahoma City, Oklahoma
  - Providence Multiple Sclerosis Center-Site Number:8400020, Portland, Oregon
  - University of Texas Southwestern Medical Center-Site Number:8400077, Dallas, Texas
  - Multiple Sclerosis Center, Swedish Neuroscience Institute-Site Number:8400121, Seattle, Washington
- Investigational Site Number :0400004, Linz, Austria
- Belarus (2):
  - Investigational Site Number :1120005, Vitebsk
  - Investigational Site Number :1120004, Vitebsk
- Bulgaria (7):
  - Investigational Site Number :1000002, Pleven
  - Investigational Site Number :1000005, Plovdiv
  - Investigational Site Number :1000004, Sofia
  - Investigational Site Number :1000008, Sofia
  - Investigational Site Number :1000001, Sofia
  - Investigational Site Number :1000006, Sofia
  - Investigational Site Number :1000009, Sofia
- Canada (4):
  - Investigational Site Number :1240016, Vancouver, British Columbia
  - Investigational Site Number :1240003, Ottawa, Ontario
  - Investigational Site Number :1240013, Toronto, Ontario
  - Investigational Site Number :1240006, Gatineau, Quebec
- China (28):
  - Investigational Site Number :1560022, Baotou
  - Investigational Site Number :1560006, Beijing
  - Investigational Site Number :1560010, Beijing
  - Investigational Site Number :1560012, Beijing
  - Investigational Site Number :1560023, Beijing
  - Investigational Site Number :1560001, Beijing
  - Investigational Site Number :1560009, Beijing
  - Investigational Site Number :1560025, Beijing
  - Investigational Site Number :1560021, Beijing
  - Investigational Site Number :1560004, Changchun
  - Investigational Site Number :1560015, Changsha
  - Investigational Site Number :1560005, Chengdu
  - Investigational Site Number :1560019, Chongqing
  - Investigational Site Number :1560035, Fuzhou
  - Investigational Site Number :1560016, Guangzhou
  - Investigational Site Number :1560028, Guangzhou
  - Investigational Site Number :1560002, Guangzhou
  - Investigational Site Number :1560027, Hohhot
  - Investigational Site Number :1560044, Nanjing
  - Investigational Site Number :1560042, Nanjing
  - Investigational Site Number :1560003, Shanghai
  - Investigational Site Number :1560018, Shenyang
  - Investigational Site Number :1560014, Shijiazhuang
  - Investigational Site Number :1560008, Taiyuan
  - Investigational Site Number :1560020, Tianjin
  - Investigational Site Number :1560011, Wuhan
  - Investigational Site Number :1560017, Xi'an
  - Investigational Site Number :1560033, Yinchuan
- Czechia (4):
  - Investigational Site Number :2030004, Hradec Králové
  - Investigational Site Number :2030009, Pardubice
  - Investigational Site Number :2030003, Teplice
  - Investigational Site Number :2030007, Zlín
- Denmark (2):
  - Investigational Site Number :2080001, Esbjerg
  - Investigational Site Number :2080005, Holstebro
- Estonia (2):
  - Investigational Site Number :2330001, Tallinn
  - Investigational Site Number :2330002, Tartu
- Finland (3):
  - Investigational Site Number :2460003, Helsinki
  - Investigational Site Number :2460001, Tampere
  - Investigational Site Number :2460002, Turku
- Germany (6):
  - Investigational Site Number :2760001, Dresden
  - Investigational Site Number :2760019, Düsseldorf
  - Investigational Site Number :2760016, Hamburg
  - Investigational Site Number :2760008, Münster
  - Investigational Site Number :2760004, Rostock
  - Investigational Site Number :2760011, Ulm
- Investigational Site Number : 3440001, Shatin, NT, Hong Kong
- Italy (14):
  - Investigational Site Number :3800002, Pozzilli, Isernia
  - Investigational Site Number :3800007, Orbassano, Torino
  - Investigational Site Number :3800011, Bergamo
  - Investigational Site Number :3800015, Catania
  - Investigational Site Number :3800012, Florence
  - Investigational Site Number :3800014, Genova
  - Investigational Site Number :3800001, Milan
  - Investigational Site Number :3800010, Milan
  - Investigational Site Number :3800003, Napoli
  - Investigational Site Number :3800006, Napoli
  - Investigational Site Number :3800008, Pavia
  - Investigational Site Number :3800005, Roma
  - Investigational Site Number :3800009, Roma
  - Investigational Site Number :3800013, Roma
- Japan (14):
  - Investigational Site Number :3920016, Chiba, Chiba
  - Investigational Site Number :3920008, Koriyama-shi, Fukushima
  - Investigational Site Number :3920012, Tsukuba, Ibaraki
  - Investigational Site Number :3920022, Morioka, Iwate
  - Investigational Site Number :3920005, Niigata, Niigata
  - Investigational Site Number :3920004, Moriguchi-shi, Osaka
  - Investigational Site Number :3920001, Osaka, Osaka
  - Investigational Site Number :3920018, Kawagoe-shi, Saitama
  - Investigational Site Number :3920014, Bunkyo-ku, Tokyo
  - Investigational Site Number :3920003, Kodaira-shi, Tokyo
  - Investigational Site Number :3920010, Ōta-ku, Tokyo
  - Investigational Site Number :3920013, Shinjuku-ku, Tokyo
  - Investigational Site Number :3920009, Ube-shi, Yamaguchi
  - Investigational Site Number :3920023, Sagamihara-shi
- Lithuania (4):
  - Investigational Site Number :4400003, Kaunas
  - Investigational Site Number :4400002, Klaipėda
  - Investigational Site Number :4400004, Šiauliai
  - Investigational Site Number :4400001, Vilnius
- Mexico (3):
  - Investigational Site Number :4840002, México
  - Investigational Site Number :4840001, México
  - Investigational Site Number :4840003, Veracruz
- Poland (8):
  - Investigational Site Number :6160008, Plewiska, Greater Poland Voivodeship
  - Investigational Site Number :6160003, Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - Investigational Site Number :6160005, Warsaw, Masovian Voivodeship
  - Investigational Site Number :6160006, Warsaw, Masovian Voivodeship
  - Investigational Site Number :6160009, Glogow Mlp., Podkarpackie Voivodeship
  - Investigational Site Number :6160002, Katowice, Silesian Voivodeship
  - Investigational Site Number :6160004, Katowice, Silesian Voivodeship
  - Investigational Site Number :6160001, Lodz
- Romania (8):
  - Investigational Site Number :6420015, Brasov
  - Investigational Site Number :6420008, Bucharest
  - Investigational Site Number :6420004, Campulung Muscel
  - Investigational Site Number :6420003, Constanța
  - Investigational Site Number :6420010, Oradea
  - Investigational Site Number :6420005, Sibiu
  - Investigational Site Number :6420001, Târgu Mureş
  - Investigational Site Number :6420002, Timișoara
- Russia (12):
  - Investigational Site Number :6430014, Krasnoyarsk
  - Investigational Site Number :6430002, Moscow
  - Investigational Site Number :6430008, Moscow
  - Investigational Site Number :6430011, Nizhny Novgorod
  - Investigational Site Number :6430003, Nizhny Novgorod
  - Investigational Site Number :6430007, Pyatigorsk
  - Investigational Site Number :6430012, Rostov-on-Don
  - Investigational Site Number :6430001, Saint Petersburg
  - Investigational Site Number :6430005, Samara
  - Investigational Site Number :6430009, Smolensk
  - Investigational Site Number :6430006, Tyumen
  - Investigational Site Number :6430004, Ufa
- Spain (8):
  - Investigational Site Number :7240003, Seville, Andalusia
  - Investigational Site Number :7240009, Barcelona, Barcelona [Barcelona]
  - Investigational Site Number :7240008, Donostia / San Sebastian, Basque Country
  - Investigational Site Number :7240001, Pozuelo de Alarcón, Madrid
  - Investigational Site Number :7240004, Córdoba
  - Investigational Site Number :7240005, Málaga
  - Investigational Site Number :7240006, Murcia
  - Investigational Site Number :7240007, Valencia
- Sweden (2):
  - Investigational Site Number :7520001, Gothenburg
  - Investigational Site Number :7520002, Stockholm
- Taiwan (5):
  - Investigational Site Number :1580007, Hsinchu
  - Investigational Site Number :1580005, Kaohsiung City
  - Investigational Site Number :1580003, Taichung
  - Investigational Site Number :1580002, Taipei
  - Investigational Site Number :1580006, Taoyuang
- Turkey (Türkiye) (10):
  - Investigational Site Number :7920005, Eskişehir
  - Investigational Site Number :7920011, Hatay
  - Investigational Site Number :7920002, Istanbul
  - Investigational Site Number :7920009, Istanbul
  - Investigational Site Number :7920007, Istanbul
  - Investigational Site Number :7920003, Istanbul
  - Investigational Site Number :7920008, Izmir
  - Investigational Site Number :7920010, Izmir
  - Investigational Site Number :7920001, Kocaeli
  - Investigational Site Number :7920006, Mersin
- Ukraine (8):
  - Investigational Site Number :8040011, Ivano-Frankivsk
  - Investigational Site Number :8040016, Kharkiv
  - Investigational Site Number :8040013, Kharkiv
  - Investigational Site Number :8040008, Kherson
  - Investigational Site Number :8040014, Kyiv
  - Investigational Site Number :8040010, Lutsk
  - Investigational Site Number :8040001, Lviv
  - Investigational Site Number :8040009, Odesa

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- [Derived] Oh J, Arnold DL, Cree BAC, Ionete C, Kim HJ, Sormani MP, Syed S, Chen Y, Maxwell CR, Benoit P, Turner TJ, Wallstroem E, Wiendl H; Tolebrutinib Phase 3 GEMINI 1 and 2 Trial Group. Tolebrutinib versus Teriflunomide in Relapsing Multiple Sclerosis. N Engl J Med. 2025 May 15;392(19):1893-1904. doi: 10.1056/NEJMoa2415985. Epub 2025 Apr 8. PMID 40202623
- See also: EFC16033 Plain language Results Summary — https://sanofi.trialsummaries.com/Study/StudyDetails?id=25237&tenant=MT_SNY_9011

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 162 sites in 24 countries. A total of 1152 participants were screened from 30-Jun-2020 to 04-Aug-2022, of which 178 were screen failures. Screen failures were mainly due to not meeting eligibility criteria.
Pre-assignment Details: A total of 974 participants were randomized in this study in a 1:1 ratio to either teriflunomide 14 milligrams (mg) or tolebrutinib 60 mg group. This was an event-driven (6-month confirmed disability worsening [CDW]) trial with a variable treatment duration (end-of-study [EOS] duration: up to approximately 48 months).
Groups:
- Teriflunomide 14 mg: Participants received teriflunomide 14 mg tablet orally once daily (QD) along with a placebo matched to tolebrutinib orally QD up to approximately 47 months.
- Tolebrutinib 60 mg: Participants received tolebrutinib 60 mg tablet orally QD along with a placebo matched to teriflunomide orally QD up to approximately 48 months.
Period: Overall Study
Arm/Group | Teriflunomide 14 mg | Tolebrutinib 60 mg
Started | 488 | 486
Completed | 415 | 409
Not Completed | 73 | 77
Not completed — Poor compliance to protocol | 2 | 4
Not completed — Withdrawal by Subject | 64 | 66
Not completed — Other | 6 | 7
Not completed — Missing study status | 1 | 0

BASELINE CHARACTERISTICS:
Population: Analysis was performed on the randomized population.
Groups:
- Teriflunomide 14 mg: Participants received teriflunomide 14 mg tablet orally QD along with a placebo matched to tolebrutinib orally QD up to approximately 47 months.
- Total: Total of all reporting groups
Arm/Group | Teriflunomide 14 mg | Tolebrutinib 60 mg | Total
Number analyzed (Participants) | 488 | 486 | 974
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.6 (9.4) | 36.8 (9.0) | 36.7 (9.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 325 | 334 | 659
  Male | 163 | 152 | 315
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 6 | 9
  Asian | 67 | 78 | 145
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 10 | 4 | 14
  White | 406 | 395 | 801
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Annualized Relapse Rate (ARR) as Assessed by Confirmed Protocol-defined Adjudicated Relapses
Description: Multiple sclerosis (MS) relapse was defined as a monophasic, acute or subacute onset of new neurological symptoms or worsening of previous neurological symptoms with an objective change on neurological examination. Symptoms were attributable to MS, lasted for >=24 hours with or without recovery, present at normal body temperature, and preceded by >=30 days of clinical stability.
Time Frame: Baseline (Day 1) to approximately 48 months
Population: The intent-to-treat (ITT) population included all randomized participants according to the intervention group allocated by the randomization, irrespective of the study intervention received.
Measure: Number (95% Confidence Interval); unit: relapses per participant year
Arm/Group | Teriflunomide 14 mg | Tolebrutinib 60 mg
Number analyzed (Participants) | 488 | 486
relapses per participant year | 0.122 [0.100 to 0.150] | 0.130 [0.108 to 0.156]
Statistical Analysis 1: Comparison: Teriflunomide 14 mg vs Tolebrutinib 60 mg; Analysis was performed using negative binomial model with number of adjudicated relapses onset between randomization date and EOS date as the response variable, treatment group, Gadolinium (Gd)-enhancing T1 lesions at baseline (presence, absence), expanded disability status scale (EDSS) strata (<4, >=4) and geographic region (United States [US], non-US) as covariates, and log transformed observation duration as the offset variable; Test type: Superiority — A hierarchical testing procedure was used to control the overall type I error; p = 0.6691, Chi-squared — Threshold for significance at 2-sided 0.05 level; Relative risk = 1.061, 95% CI 2-sided [0.808 to 1.393]

2. Secondary Outcome: Time to Onset of 6-Month Confirmed Disability Worsening as Assessed by Expanded Disability Status Scale
Description: The EDSS was a disability scale that assessed the following 7 functional domains: visual, brainstem, pyramidal [motor], cerebellar [coordination], sensory, cerebral, and bowel/bladder. The total EDSS score ranged from 0 (normal) to 10 (death due to MS), increasing in increments of 0.5 points. Higher scores indicated increased disability. Time to onset of 6-month CDW was defined as the time from randomization to the onset of a confirmed, sustained increase from baseline in EDSS score (of >=1.5 points when the baseline score was 0, of >=1.0 point when the baseline score was 0.5 to <=5.5, of >=0.5 points when the baseline EDSS score was >5.5) over at least 6 months that was not attributable to another etiology.
Time Frame: Baseline (Day 1) to approximately 48 months
Population: The ITT population included all randomized participants according to the intervention group allocated by the randomization, irrespective of the study intervention received.
Measure: Median (Full Range); unit: months
Arm/Group | Teriflunomide 14 mg | Tolebrutinib 60 mg
Number analyzed (Participants) | 488 | 486
months | 17.97 [2.9 to 33.9] | 15.38 [2.6 to 36.8]
Statistical Analysis 1: Comparison: Teriflunomide 14 mg vs Tolebrutinib 60 mg; Analysis was performed using Cox proportional-hazards model with robust variance estimation. Covariates were treatment group, Gd-enhancing T1 lesions at baseline (presence, absence), EDSS strata (<4, >=4), geographic region (US, non-US); Test type: Superiority — A hierarchical testing procedure was used to control the overall type I error; p = 0.4888, Log Rank — Derived from log-rank test with stratification of EDSS strata (<4, >=4), geographic region (US, non-US); Hazard Ratio (HR) = 0.850, 95% CI 2-sided [0.565 to 1.278]

3. Secondary Outcome: Time to Onset of 3-Month Confirmed Disability Worsening as Assessed by Expanded Disability Status Scale
Description: The EDSS was a disability scale that assessed the following 7 functional domains: visual, brainstem, pyramidal [motor], cerebellar [coordination], sensory, cerebral, and bowel/bladder. The total EDSS score ranged from 0 (normal) to 10 (death due to MS), increasing in increments of 0.5 points. Higher scores indicated increased disability. Time to onset of 3-month CDW was defined as the time from randomization to the onset of a confirmed, sustained increase from baseline in EDSS score (of >=1.5 points when the baseline score was 0, of >=1.0 point when the baseline score was 0.5 to <=5.5, of >=0.5 points when the baseline EDSS score was >5.5) over at least 3 months that was not attributable to another etiology.
Time Frame: Baseline (Day 1) to approximately 48 months
Population: as for outcome 2
Measure: Median (Full Range); unit: months
Arm/Group | Teriflunomide 14 mg | Tolebrutinib 60 mg
Number analyzed (Participants) | 488 | 486
months | 17.96 [2.9 to 39.3] | 14.93 [0.2 to 41.0]
Statistical Analysis 1: Comparison: Teriflunomide 14 mg vs Tolebrutinib 60 mg; [analysis description as in outcome 2, analysis 1]; Test type: Superiority — A hierarchical testing procedure was used to control the overall type I error; p = 0.2991, Log Rank — Derived from log-rank test with stratification of EDSS strata (<4, >=4), geographic region (US, non-US); Hazard Ratio (HR) = 0.819, 95% CI 2-sided [0.582 to 1.151]

4. Secondary Outcome: Mean Number of New and/or Enlarging T2-Hyperintense Lesions Per Year
Description: Magnetic resonance imaging (MRI) of the brain was performed to identify number of new and/or enlarging T2-hyperintense lesions defined as the sum of the individual number of new and/or enlarging T2 lesions starting from baseline up to and including the EOS visit.
Time Frame: Baseline (Day 1) to approximately 48 months
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: number of new and or enlarging T2lesions
Arm/Group | Teriflunomide 14 mg | Tolebrutinib 60 mg
Number analyzed (Participants) | 488 | 486
number of new and or enlarging T2lesions | 5.175 [4.447 to 6.024] | 5.611 [4.826 to 6.524]
Statistical Analysis 1: Comparison: Teriflunomide 14 mg vs Tolebrutinib 60 mg; Analysis was performed using negative binomial model with the number of new and/or enlarging T2-hyperintense lesions between randomization date and EOS date as the response variable, treatment group, baseline T2-hyperintense lesion count, EDSS strata (<4, >=4) and geographic region (US, non-US) as covariates, and log transformed observation duration as the offset variable; Test type: Superiority — A hierarchical testing procedure was used to control the overall type I error; p = 0.4575, Chi-squared; Relative risk = 1.084, 95% CI 2-sided [0.876 to 1.342]

5. Secondary Outcome: Mean Number of New Gadolinium-Enhancing T1-Hyperintense Lesions Per Scan
Description: MRI of the brain was performed to identify number of new Gd-enhancing T1-hyperintense lesions defined as the sum of the individual number of new Gd- enhancing T1-hyperintense lesions starting from baseline up to and including the EOS visit.
Time Frame: Baseline (Day 1) to approximately 48 months
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: number of new Gd-enhancing T1 lesions
Arm/Group | Teriflunomide 14 mg | Tolebrutinib 60 mg
Number analyzed (Participants) | 488 | 486
number of new Gd-enhancing T1 lesions | 0.285 [0.221 to 0.367] | 0.530 [0.439 to 0.641]
Statistical Analysis 1: Comparison: Teriflunomide 14 mg vs Tolebrutinib 60 mg; Analysis was performed using negative binomial model with the number of new Gd-enhancing T1-hyperintense lesions between randomization date and EOS date as the response variable, treatment group, Gd-enhancing T1 lesions at baseline (presence, absence), EDSS strata (<4, >=4) and geographic region (US, non-US) as covariates, and log transformed number of MRI scans as the offset variable; Test type: Superiority — A hierarchical testing procedure was used to control the overall type I error; p = 0.0001, Chi-squared; Relative risk = 1.860, 95% CI 2-sided [1.358 to 2.548]

6. Secondary Outcome: Change From Baseline in Cognitive Function as Assessed by the Symbol Digit Modalities Test (SDMT) at EOS
Description: The SDMT was used to assess processing speed, divided attention, visual scanning, tracking and motor speed. It involved a simple substitution task using a reference key. The number of correct substitutions and number of items completed within a 90 second interval (maximum 110 seconds) were recorded. A decrease of 4 points from baseline on the SDMT was considered meaningful worsening. The score was the number of correctly coded items from 0-110 in 90 seconds; higher scores indicating a better outcome. Baseline was defined as the last available value prior to the first dose of study intervention.
Time Frame: Baseline (Day 1) to EOS (up to approximately 48 months)
Population: The ITT population included all randomized participants according to the intervention group allocated by the randomization, irrespective of the study intervention received. Only participants with data collected at specified timepoints are reported.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Teriflunomide 14 mg | Tolebrutinib 60 mg
Number analyzed (Participants) | 396 | 393
score on a scale | 0.329 (0.0318) | 0.364 (0.0318)
Statistical Analysis 1: Comparison: Teriflunomide 14 mg vs Tolebrutinib 60 mg; Covariates in the mixed-effect model with repeated measures (MMRM) were treatment group, EDSS strata (<4, >=4), geographic region (US, non-US), visit, treatment by visit interaction, baseline value, and baseline value-by-visit interaction; Test type: Superiority — A hierarchical testing procedure was used to control the overall type I error; p = 0.4320, MMRM; Least square (LS) mean difference = 0.035, 95% CI 2-sided [-0.053 to 0.124]

7. Secondary Outcome: Change From Baseline in Cognitive Function as Assessed by the California Verbal Learning Test Second Edition (CVLT-II) at EOS
Description: The CVLT-II was a verbal learning and memory test consisting of recall and recognition of a list of 16 words. For each assessment, 5 trials were completed. Total Correct Recall Trials 1-5 was scaled to a normalized T-score metric, which had a mean of 50 and standard deviation of 10, the maximum possible score was 80 and a minimum was 0. Higher values indicated improved cognitive function. Baseline was defined as the last available value prior to the first dose of study intervention.
Time Frame: Baseline (Day 1) to EOS (up to approximately 48 months)
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: T-score
Arm/Group | Teriflunomide 14 mg | Tolebrutinib 60 mg
Number analyzed (Participants) | 391 | 390
T-score | 15.827 (0.7241) | 17.700 (0.7236)
Statistical Analysis 1: Comparison: Teriflunomide 14 mg vs Tolebrutinib 60 mg; Covariates in the MMRM were treatment group, EDSS strata (<4, >=4), geographic region (US, non-US), visit, treatment by visit interaction, baseline value, and baseline value-by-visit interaction; Test type: Superiority — A hierarchical testing procedure was used to control the overall type I error; p = 0.0675, MMRM; LS mean difference = 1.873, 95% CI 2-sided [-0.135 to 3.880]

8. Secondary Outcome: Time to Onset of 6-Month Confirmed Disability Improvement (CDI) as Assessed by Expanded Disability Status Scale
Description: The EDSS was a disability scale that assessed the following 7 functional domains: visual, brainstem, pyramidal [motor], cerebellar [coordination], sensory, cerebral, and bowel/bladder. The total EDSS score ranged from 0 (normal) to 10 (death due to MS), increasing in increments of 0.5 points. Higher scores indicated increased disability. CDI was defined as a decrease of >=1 point from baseline in the EDSS score lasting at least 6 months.
Time Frame: Baseline (Day 1) to approximately 48 months
Population: as for outcome 2
Measure: Median (Full Range); unit: months
Arm/Group | Teriflunomide 14 mg | Tolebrutinib 60 mg
Number analyzed (Participants) | 488 | 486
months | 12.04 [2.8 to 37.1] | 11.82 [2.8 to 33.0]
Statistical Analysis 1: Comparison: Teriflunomide 14 mg vs Tolebrutinib 60 mg; [analysis description as in outcome 2, analysis 1]; Test type: Superiority — A hierarchical testing procedure was used to control the overall type I error; p = 0.3594, Log Rank — Derived from log-rank test with stratification of EDSS strata (<4, >=4), geographic region (US, non-US); Hazard Ratio (HR) = 0.831, 95% CI 2-sided [0.554 to 1.245]

9. Secondary Outcome: Percent Change in Brain Volume Loss at EOS Compared to Month 6
Description: MRI of the brain was performed at the specified timepoints to detect the changes in brain volume loss.
Time Frame: Month 6 to EOS (up to approximately 48 months)
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Teriflunomide 14 mg | Tolebrutinib 60 mg
Number analyzed (Participants) | 346 | 351
percent change | -0.884 (0.0368) | -0.688 (0.0369)
Statistical Analysis 1: Comparison: Teriflunomide 14 mg vs Tolebrutinib 60 mg; Covariates in the MMRM were treatment group, EDSS strata (<4, >=4), geographic region (US, non-US), visit, treatment by visit interaction, cube root transformed Month 6 brain volume, and cube root transformed Month 6 brain volume-by-visit interaction; Test type: Superiority — A hierarchical testing procedure was used to control the overall type I error; p = 0.0002, MMRM; LS mean difference = 0.196, 95% CI 2-sided [0.093 to 0.298]

10. Secondary Outcome: Change From Baseline in Multiple Sclerosis Quality of Life 54 (MSQoL-54) Questionnaire Score at EOS
Description: MSQoL-54 was standardized instrument comprising generic and MS-specific items. This 54-item instrument generated 12 subscales and 2 single-item measures (satisfaction with sexual function [1 item]; change in health [1 item]). 12 subscales were: a: physical health (10 items), b: health perceptions (5 items), c: energy (5 items), d: role limit physical (4 items), e: sexual function (4 items), f: pain (3 items), g: social function (3 items), h: health distress (4 items), i: overall quality of life (2 items), j: emotional well-being (5 items), k: role limitations emotional (3 items) and l: cognitive function (4 items). Physical and mental health composite score were calculated as weighted sum of 'a to h' and 'i to l' subscales respectively. Each composite score was transformed linearly to common 0 (worst) to 100 (best) score range; higher score indicated improved quality of life. Baseline was defined as last available value prior to first dose of study intervention.
Time Frame: Baseline (Day 1) to EOS (up to approximately 48 months)
Population: The ITT population included all randomized participants according to the intervention group allocated by the randomization, irrespective of the study intervention received. Only participants with data collected at specified timepoints for the specified categories are reported.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Teriflunomide 14 mg | Tolebrutinib 60 mg
Number analyzed (Participants) | 400 | 399
score on a scale
  Physical health composite score: number analyzed (Participants) | 393 | 394
  Physical health composite score | -2.468 (0.7014) | -0.460 (0.7021)
  Mental health composite score | -2.070 (0.8346) | -0.729 (0.8359)

11. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs), Treatment-emergent Serious Adverse Events (TESAEs), TEAEs Leading to Permanent Study Intervention Discontinuation and Treatment-emergent Adverse Events of Special Interest (AESIs)
Description: An AE was any untoward medical occurrence in a participant or clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. SAE was any untoward medical occurrence that at any dose: resulted in death, was life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent disability/incapacity, was a congenital anomaly/birth defect or was an important medical event. An AESI was an AE (serious or nonserious) of scientific and medical concern specific to the Sponsor's product or program for which ongoing monitoring and immediate notification by the Investigator to the Sponsor was required. TEAEs were defined as AEs that developed, worsened or became serious during the TE period.
Time Frame: From first dose of study intervention (Day 1) up to the earliest of either 10 days post last dose, death or last contact; up to approximately 48 months
Population: The safety population included all randomized participants exposed to the study intervention, regardless of the amount of exposure, analyzed according to the intervention actually received.
Measure: Count of Participants; unit: Participants
Arm/Group | Teriflunomide 14 mg | Tolebrutinib 60 mg
Number analyzed (Participants) | 488 | 486
Participants
  TEAEs | 423 | 407
  TESAEs | 40 | 42
  TEAEs leading to permanent study intervention discontinuation | 24 | 23
  TEAESIs | 57 | 53

12. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of Tolebrutinib and M2 Metabolite
Description: Blood samples were collected at specified timepoints to assess Cmax of tolebrutinib and M2 metabolite using population pharmacokinetic (PK) model.
Time Frame: 30-90 minutes post-dose at Months 6, 9, and 12 and 2.5-5 hours post-dose at Months 6 and 12
Population: The PK population included all participants in the safety population with at least 1 non-missing PK sample after first dose of the study intervention. Only participants with data collected at specified timepoints are reported.
Measure: Mean (Standard Deviation); unit: nanogram/milliliter (ng/mL)
Arm/Group | Tolebrutinib 60 mg
Number analyzed (Participants) | 444
nanogram/milliliter (ng/mL)
  Tolebrutinib | 12.0 (7.75)
  M2 Metabolite | 28.3 (15.8)

13. Secondary Outcome: Time to Maximum Observed Plasma Concentration (Tmax) of Tolebrutinib and M2 Metabolite
Description: Blood samples were collected at specified timepoints to assess Tmax of tolebrutinib and M2 metabolite using population PK model.
Time Frame: 30-90 minutes post-dose at Months 6, 9, and 12 and 2.5-5 hours post-dose at Months 6 and 12
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: hour (h)
Arm/Group | Tolebrutinib 60 mg
Number analyzed (Participants) | 444
hour (h)
  Tolebrutinib | 1.28 (0.513)
  M2 Metabolite | 1.40 (0.508)

14. Secondary Outcome: Area Under the Plasma Concentration-time Curve Over the Last 24-hours Dosing Interval (AUC0-24) of Tolebrutinib and M2 Metabolite
Description: Blood samples were collected at specified timepoints to assess AUC0-24 of tolebrutinib and M2 metabolite using population PK model.
Time Frame: 30-90 minutes post-dose at Months 6, 9, and 12 and 2.5-5 hours post-dose at Months 6 and 12
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Tolebrutinib 60 mg
Number analyzed (Participants) | 444
ng*h/mL
  Tolebrutinib | 30.5 (18.2)
  M2 Metabolite | 76.7 (44.1)

15. Secondary Outcome: Change From Baseline in Plasma Neurofilament Light Chain (NfL) and Serum Chitinase-3 Like Protein-1 (Chi3L1) Levels at EOS
Description: Blood samples were collected at specified timepoints to assess change from baseline in NfL and Chi3L1. Baseline was defined as the last available value prior to the first dose of study intervention.
Time Frame: Baseline (Day 1) to EOS (up to approximately 48 months)
Population: The safety population included all randomized participants exposed to the study intervention, regardless of the amount of exposure, analyzed according to the intervention actually received. Only participants with data collected at specified timepoints for the specified categories are reported.
Measure: Median (Inter-Quartile Range); unit: picogram/mL
Arm/Group | Teriflunomide 14 mg | Tolebrutinib 60 mg
Number analyzed (Participants) | 344 | 350
picogram/mL
  NfL: number analyzed (Participants) | 294 | 296
  NfL | -1.665 [-6.100 to 0.830] | -0.325 [-3.505 to 2.220]
  Chi3L1 | 1017.100 [-4494.850 to 7672.450] | 1572.250 [-2582.000 to 6356.600]

16. Secondary Outcome: Change From Baseline in Cluster of Differentiation (CD)19+ B Cells at EOS
Description: Blood samples were collected at specified timepoints to assess change from baseline in CD19+ B cells. Baseline was defined as the last available value prior to the first dose of study intervention.
Time Frame: Baseline (Day 1) to EOS (up to approximately 48 months)
Population: The safety population included all randomized participants exposed to the study intervention, regardless of the amount of exposure, analyzed according to the intervention actually received. Only participants with data collected at specified timepoints are reported.
Measure: Median (Inter-Quartile Range); unit: cells/microliter
Arm/Group | Teriflunomide 14 mg | Tolebrutinib 60 mg
Number analyzed (Participants) | 95 | 100
cells/microliter | -45.000 [-81.000 to -5.000] | -60.500 [-97.500 to -28.500]

17. Secondary Outcome: Change From Baseline in Serum Immunoglobulin (Ig) Levels at EOS
Description: Blood samples were collected at specified timepoints to assess change from baseline in IgG and IgM levels. Baseline was defined as the last available value prior to the first dose of study intervention.
Time Frame: Baseline (Day 1) to EOS (up to approximately 48 months)
Population: as for outcome 15
Measure: Median (Inter-Quartile Range); unit: gram/liter
Arm/Group | Teriflunomide 14 mg | Tolebrutinib 60 mg
Number analyzed (Participants) | 263 | 266
gram/liter
  IgG: number analyzed (Participants) | 261 | 266
  IgG | -0.660 [-1.460 to 0.150] | 0.235 [-0.500 to 1.020]
  IgM: number analyzed (Participants) | 263 | 263
  IgM | -0.150 [-0.330 to -0.030] | -0.340 [-0.520 to -0.190]

ADVERSE EVENTS:
Time Frame: From first dose of study intervention (Day 1) up to the earliest of either 10 days post last dose, death or last contact; up to approximately 48 months. Deaths were collected from baseline (Day 1) up to end of follow-up, approximately 48 months.
Description: Analysis was performed on the safety population. This was an event-driven (6-month CDW) trial with a variable treatment duration (EOS duration: up to approximately 48 months).
Arm/Group | Teriflunomide 14 mg | Tolebrutinib 60 mg
All-Cause Mortality (participants affected / at risk) | 0/488 | 0/486
Serious Adverse Events (participants affected / at risk) | 40/488 | 42/486
Other Adverse Events (participants affected / at risk) | 321/488 | 296/486
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Teriflunomide 14 mg (N=488) | Tolebrutinib 60 mg (N=486)
Appendicitis (Infections and infestations) | 0 (0) | 2 (2)
Covid-19 (Infections and infestations) | 1 (1) | 1 (1)
Covid-19 Pneumonia (Infections and infestations) | 2 (2) | 4 (4)
Chronic Sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Chronic Tonsillitis (Infections and infestations) | 0 (0) | 1 (1)
Cystitis (Infections and infestations) | 1 (1) | 0 (0)
Enteritis Infectious (Infections and infestations) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 1 (1) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 1 (1)
Pyelonephritis Acute (Infections and infestations) | 0 (0) | 1 (1)
Respiratory Tract Chlamydial Infection (Infections and infestations) | 1 (1) | 0 (0)
Salpingo-Oophoritis (Infections and infestations) | 0 (0) | 1 (1)
Systemic Viral Infection (Infections and infestations) | 1 (1) | 0 (0)
Viral Upper Respiratory Tract Infection (Infections and infestations) | 1 (1) | 0 (0)
Adenocarcinoma Of Colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Benign Bone Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Benign Ovarian Tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Bladder Transitional Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Breast Cancer Stage Ii (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Invasive Breast Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Renal Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Soft Tissue Sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Uterine Leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Thinking Abnormal (Psychiatric disorders) | 1 (1) | 0 (0)
Central Nervous System Lesion (Nervous system disorders) | 1 (1) | 0 (0)
Epilepsy (Nervous system disorders) | 0 (0) | 1 (1)
Multiple Sclerosis Relapse (Nervous system disorders) | 5 (6) | 3 (3)
Optic Neuritis (Nervous system disorders) | 1 (1) | 0 (0)
Sciatica (Nervous system disorders) | 2 (2) | 0 (0)
Status Epilepticus (Nervous system disorders) | 0 (0) | 1 (1)
Diplopia (Eye disorders) | 1 (1) | 0 (0)
Vision Blurred (Eye disorders) | 1 (1) | 0 (0)
Visual Field Defect (Eye disorders) | 1 (1) | 0 (0)
Visual Impairment (Eye disorders) | 1 (1) | 1 (1)
Supraventricular Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Hypertensive Crisis (Vascular disorders) | 1 (1) | 0 (0)
Varicose Vein (Vascular disorders) | 0 (0) | 1 (1)
Nasal Septum Deviation (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Abdominal Pain Upper (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Duodenal Ulcer Haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Epulis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Food Poisoning (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal Disorder (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal Erosion (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis Acute (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Bile Duct Stone (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholecystitis Chronic (Hepatobiliary disorders) | 1 (1) | 0 (0)
Drug-Induced Liver Injury (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatic Function Abnormal (Hepatobiliary disorders) | 1 (1) | 0 (0)
Erythema Multiforme (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Intervertebral Disc Protrusion (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Rotator Cuff Syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Abortion Spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 2 (2)
Endometriosis (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Intermenstrual Bleeding (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Uterine Haemorrhage (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Alanine Aminotransferase Increased (Investigations) | 1 (1) | 0 (0)
Blood Pressure Increased (Investigations) | 1 (1) | 0 (0)
Transaminases Increased (Investigations) | 0 (0) | 1 (1)
Burns Second Degree (Injury, poisoning and procedural complications) | 0 (0) | 1 (2)
Femur Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Forearm Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hyphaema (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Joint Dislocation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Limb Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Meniscus Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Multiple Fractures (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Patella Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Rib Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Teriflunomide 14 mg (N=488) | Tolebrutinib 60 mg (N=486)
Covid-19 (Infections and infestations) | 135 (150) | 117 (133)
Influenza (Infections and infestations) | 26 (35) | 19 (24)
Nasopharyngitis (Infections and infestations) | 41 (61) | 59 (88)
Upper Respiratory Tract Infection (Infections and infestations) | 46 (65) | 46 (69)
Urinary Tract Infection (Infections and infestations) | 27 (32) | 34 (45)
Viral Upper Respiratory Tract Infection (Infections and infestations) | 34 (48) | 31 (54)
Neutropenia (Blood and lymphatic system disorders) | 58 (93) | 14 (22)
Depression (Psychiatric disorders) | 27 (27) | 11 (11)
Headache (Nervous system disorders) | 44 (62) | 56 (100)
Hypertension (Vascular disorders) | 27 (28) | 16 (19)
Diarrhoea (Gastrointestinal disorders) | 36 (50) | 22 (24)
Alopecia (Skin and subcutaneous tissue disorders) | 73 (75) | 36 (36)
Arthralgia (Musculoskeletal and connective tissue disorders) | 27 (31) | 18 (25)
Back Pain (Musculoskeletal and connective tissue disorders) | 30 (34) | 31 (35)
Alanine Aminotransferase Increased (Investigations) | 40 (43) | 23 (26)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor supports publication of clinical trial results but may request that investigators temporarily delay or alter publications in order to protect proprietary information. The Sponsor may also require that the results of multicenter studies be published only in their entirety and not as individual site data.

DOCUMENTS (2):
  • Study Protocol (2023-12-20): https://cdn.clinicaltrials.gov/large-docs/78/NCT04410978/Prot_000.pdf
  • Statistical Analysis Plan (2024-07-10): https://cdn.clinicaltrials.gov/large-docs/78/NCT04410978/SAP_001.pdf